CLINICAL TRIAL: NCT01187836
Title: A Randomized, Double-Blind, Placebo-Controlled, Adaptive, Ascending Dose-Titration Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Invasive Hemodynamics of TRV120027 in Patients With Stable Heart Failure
Brief Title: Study to Evaluate the Effects of TRV120027 in Patients With Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP120027.2001; 2010-020376-37 (EudraCT Number)
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sar-Arg-Val-Tyr-Ile-His-Pro-Ala-OH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- TRV120027 (Experimental)
  Interventions: Drug: TRV120027
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRV120027 — Dose range (starting at 0.1 mcg/kg/min) of TRV120027 administered for 14 hours.
  Arms: TRV120027
Drug: Placebo — Placebo administered for 14 hours.
  Arms: Placebo

SUMMARY:
In this study, TRV120027 (or a placebo) intravenous infusion will be given to people with heart failure to learn about the effects of TRV120027. The results of this study will help choose the proper range of TRV120027 doses to use in future research studies involving patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congestive heart failure made at least 3 months prior to screening
* NYHA Class III or IV heart failure, ejection fraction </= 35% and , and in the opinion of the investigator, right-heart catheterization is clinically indicated.
* Baseline mean PCWP >/= 20 mmHg
* Systolic blood pressure at screening must be >/= 100 mmHg. Heart rate at screening must be </= 90 bpm.

Exclusion Criteria:

* Any significant disease or condition that would interfere with the interpretation of safety or efficacy in this study as determined by the Investigator based on medical history, physical examination or laboratory tests.
* Significant valve disease
* Current signs or symptoms of acute myocardial ischemia or acute coronary syndrome (ACS) or coronary revascularization in the past 3 months.
* Sustained or uncontrolled ventricular arrhythmia. Inclusion of patients with atrial fibrillation with a heart rate ≤ 90 bpm is permitted.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary Capillary Wedge Pressure (PCWP) | Multiple time points during 14 hr infusion and during 4 hr period after end of infusion
  The effect of TRV120027 on pulmonary capillary wedge pressure will be compared to baseline and to placebo at multiple measurement time points during the 14 hour infusion and for 4 hours after discontinuation of the infusion.
Safety and Tolerability | Multiple time points during 14 hr infusion and during 4 hr period after end of infusion, and follow-up (Day 7, Day 30)
  Safety and tolerability will be assessed qualitatively by evaluating adverse events, clinical laboratories, ECGs, cardiac telemetry and vital signs at multiple measurement time points during the 14 hour infusion and for 4 hours after discontinuation of the infusion. Follow-up assessments for adverse events at Day 7 and Day 30 will be conducted.

SECONDARY OUTCOMES:
Pharmacokinetics of TRV120027 | Multiple time points during 14 hr infusion and during 4 hr period after end of infusion
  PK samples will be collected at multiple time points during the 14 hour infusion and 4 hour washout periods.
Additional Hemodynamics | Multiple time points during 14 hr infusion and during 4 hr period after end of infusion
  Additional hemodynamic variables (for example, right atrial pressure, pulmonary arterial pressure and cardiac output) will be compared to baseline and to placebo at multiple measurement time points during the 14 hour infusion and for 4 hours after discontinuation of the infusion.
Laboratory Evaluations | Multiple time points during 14 hr infusion and during 4 hr period after end of infusion, and follow-up (Day 7)
  Biomarkers of renal function and neurohormonal activation will be assessed at multiple measurement time points during the 14 hour infusion and for 4 hours after discontinuation of the infusion, and again at follow-up Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: David G Soergel, M.D., Study Director — Trevena Inc.
Locations (9):
- United States (4):
  - Miami, Florida
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Utah, Salt Lake City, Utah
- Czechia (3):
  - CZ05, Brno
  - CZ04, Olomouc
  - CZ06, Prague
- Poland (2):
  - PL01, Warsaw
  - PL05, Wroclaw